CLINICAL TRIAL: NCT02371174
Title: An Observational Post-Marketing Surveillance Study on the Status and Factors for the Development of Peripheral Neuropathy in Patients With HER2-Negative Inoperable or Recurrent Breast Cancer in Japan.
Brief Title: Post-Marketing Surveillance Study of Eribulin on the Status and Factors for the Development of Peripheral Neuropathy in Japan.
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: HAL02T
Record Dates: First submitted 2014-11-21; First posted 2015-02-25 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer
Keywords: HER2-Negative Inoperable or Recurrent Breast Cancer; Japan; Eribulin Mesylate
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HALAVEN treatment group of primary or secondary chemotherapy: Patients with HER2-negative recurrent breast cancer who have received 0 or 1 chemotherapy regimen for recurrent breast cancer.
- HALAVEN treatment group of tertiary or later chemotherapy: Patients with HER2-negative inoperable or recurrent breast cancer who have received 2 or more chemotherapy regimens for inoperable or recurrent breast cancer.

SUMMARY:
The primary objective of the study is to clarify factors affecting the incidence of peripheral neuropathy in patients treated with HALAVEN. A total of 590 patients will be enrolled in this study with 295 patients in the treatment group of primary or secondary chemotherapy and 295 patients in the treatment group of tertiary or later chemotherapy.

ELIGIBILITY:
Inclusion criteria:

Patients with HER2-negative inoperable or recurrent breast cancer.

Exclusion criteria:

Patients with high-grade bone marrow depression (absolute neutrophil count less than 1,000 /mm^3, absolute platelet count less than 75,000 /mm^3).

Patients with a history of hypersensitivity to the ingredients of HALAVEN. Women who are pregnant or may be pregnant. Patients with a history of use of HALAVEN.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HER2-negative subjects who are treated with HALAVEN for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-01-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Baseline and up to 2 years after the initial dose of HALAVEN
Number of participants with peripheral neuropathy | Baseline, and every two months after the initial dose of HALAVEN up to 2 years
  Common Terminology Criteria for Adverse Events (CTCAE) grade of peripheral neuropathy is assessed at baseline, and every two months after the initial dose of HALAVEN up to 2 years.
Number of participants with adverse drug reactions | Baseline and up to 2 years after the initial dose of HALAVEN
Time to onset of peripheral neuropathy | Baseline and up to 2 years after the initial dose of HALAVEN
Time to resolution of peripheral neuropathy | Baseline and up to 2 years after the initial dose of HALAVEN

SECONDARY OUTCOMES:
Overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

REFERENCES:
- [Derived] Tanabe Y, Inoue K, Takahashi M, Mukai H, Yamanaka T, Egawa C, Uchida Y, Higashibeppu Y, Sakata Y, Sugawara M, Tsurutani J. Prognosis of Invasive Lobular Carcinoma and Effectiveness of Eribulin in Clinical Practice: A Post Hoc Analysis of a 2-Year Post-Marketing Surveillance. Asia Pac J Clin Oncol. 2025 Dec;21(6):623-630. doi: 10.1111/ajco.14189. Epub 2025 May 22. PMID 40404608